CLINICAL TRIAL: NCT06877546
Title: Photodynamic Treatment as Part of Oral Healthcare on Persons With Sjögren's Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: Metropolia University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PhoSS
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Sjogren Syndrome; Xerostomia
Keywords: Sjögren's syndrome; xerostomia; aPDT; antibacterial; photodynamic therapy; photobiomodulation
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumoral® Treatment (Experimental): Lumoral® Treatment is an adjunctive treatment to normal oral hygiene routines
  Interventions: Device: Lumoral treatment

INTERVENTIONS:
Device: Lumoral treatment — Lumoral® Treatment devices are handed over to study participants on the first visit. The treatment is performed first at the clinic under supervision by the researchers. Treatment is then repeated at home twice a week for 12 weeks.
  The treatment is started by dissolving one 7 mg Lumorinse® oral tablet in 30 ml amount of pure water. The tablet dissolves in water in one minute, after which the mouthwash is poured into the mouth and swished for 60 seconds. The indocyanine green in the mouthwash adheres to the plaque surface in the teeth and gum line. The mouthwash is then spat out and the mouthpiece of the Lumoral® Treatment device is inserted into the mouth and a light is activated. After 10 minutes, the device turns itself off, after which the mouthpiece is removed from the mouth. Normal oral hygiene routines will then be performed.

SUMMARY:
This thesis study will investigate whether the regular use of antibacterial photodynamic therapy can alleviate dry mouth symptoms in patients with Sjogren's syndrome and thus be a potential addition to regular oral self-care habits that promote and maintain oral health.

DETAILED DESCRIPTION:
Sjogren's syndrome is a chronic autoimmune disease that has a holistic impact on a patient's health. The most significant consequence in terms of oral health is the destruction of the salivary glands by the autoimmune reaction, leading to salivary gland failure and consequently dry mouth with reduced saliva secretion. Decreased saliva secretion predisposes to a number of oral health problems, and patients with Sjogren's syndrome are therefore at risk for conditions such as caries and periodontitis, an inflammatory periodontal disease. Regular visits to an oral health professional and good oral hygiene and eating habits and habits promote and maintain oral health. Treatments for dry mouth symptoms associated with Sjogren's syndrome aim to relieve oral symptoms by preserving, replacing and stimulating salivary gland secretion in ways that relieve local inflammation.

Regular home-use of specially designed antibacterial photodynamic therapy device in addition to standard oral self-care has been shown to destroy oral disease-causing bacteria in a way that bacteria cannot develop resistance to. In addition, the treatment method also stimulates saliva production through photobiomodulation. The aim of our study is therefore to investigate, by means of a clinical measurement, whether the regular use of the antibacterial photodynamic therapy device as part of oral self-care can have an effect on the amount of stimulated saliva secretion of a patient with Sjogren's syndrome during the ten-week study period. The aim is also to describe, by means of a questionnaire measuring the subjective symptoms of dry mouth, whether the treatment has an effect on the frequency of the typical symptoms of xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* Adult (minimum 18 years of age) person with Sjogren's syndrome, with dry mouth symptoms but some saliva secretion.
* Otherwise perceived health good, primary Sjögren's syndrome patient.
* No need for antibiotic prophylaxis at the time of a limited oral examination.
* Signed written informed consent.
* Subject's co-operation allows participation in the study.

Exclusion Criteria:

* Pregnancy and/or breastfeeding.
* Fungal infection in the mouth
* Poor oral health, such as caries lesions or advanced periodontitis.
* Fixed dentures, or orthodontics.
* No saliva secretion.
* Bisphosphonate drugs, multiple (more than two) medications in use.
* Participation in other oral health research at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-05-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Stimulated saliva | 3 months
  Measurement of stimulated saliva is performed at the baseline and study end visits. On both visits, the stimulated saliva is measured twice: before and after the investigational device use.
  Stimulated saliva production is measured in a frontal, sitting, or semi-sitting position by having the patient chew a piece of paraffin, for example, for one minute. During this time, the saliva is swallowed. The patient then continues to chew for five minutes, during which time the saliva accumulated in the mouth is drained into a measuring cup.
  The volume of stimulated saliva is measured in milliliters. The measurements will be analyzed using quantitive methods.

SECONDARY OUTCOMES:
Subjective dry mouth (xerostomia) follow-up | 3 months
  Xerostomia questionnaire.
  Study subjects are asked to fill in a questionnaire at the study end visit to determine the frequency of xerostomia symptoms during the 3-month study period. The questionnaire is designed to ask a set of pre-set questions, which are answered on a 5-point Likert scale (1, not at all true - 5, completely true).

CONTACTS AND LOCATIONS:
Overall Officials: Saila Pakarinen, DDS, Principal Investigator — Metropolia University of Applied Sciences
Locations (1):
- Metropolia University of applied sciences, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrandez-Pujante A, Pons-Fuster E, Lopez-Jornet P. Efficacy of Photobiomodulation in Reducing Symptomatology and Improving the Quality of Life in Patients with Xerostomia and Hyposalivation: A Randomized Controlled Trial. J Clin Med. 2022 Jun 14;11(12):3414. doi: 10.3390/jcm11123414. PMID 35743485
- [Background] Jao Y, Ding SJ, Chen CC. Antimicrobial photodynamic therapy for the treatment of oral infections: A systematic review. J Dent Sci. 2023 Oct;18(4):1453-1466. doi: 10.1016/j.jds.2023.07.002. Epub 2023 Jul 11. PMID 37799910
- [Background] Lahteenmaki H, Patila T, Raisanen IT, Kankuri E, Tervahartiala T, Sorsa T. Repeated Home-Applied Dual-Light Antibacterial Photodynamic Therapy Can Reduce Plaque Burden, Inflammation, and aMMP-8 in Peri-Implant Disease-A Pilot Study. Curr Issues Mol Biol. 2022 Mar 8;44(3):1273-1283. doi: 10.3390/cimb44030085. PMID 35723308
- [Background] Negrini S, Emmi G, Greco M, Borro M, Sardanelli F, Murdaca G, Indiveri F, Puppo F. Sjogren's syndrome: a systemic autoimmune disease. Clin Exp Med. 2022 Feb;22(1):9-25. doi: 10.1007/s10238-021-00728-6. Epub 2021 Jun 7. PMID 34100160
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Pakarinen S, Saarela RKT, Valimaa H, Heikkinen AM, Kankuri E, Noponen M, Alapulli H, Tervahartiala T, Raisanen IT, Sorsa T, Patila T. Home-Applied Dual-Light Photodynamic Therapy in the Treatment of Stable Chronic Periodontitis (HOPE-CP)-Three-Month Interim Results. Dent J (Basel). 2022 Nov 2;10(11):206. doi: 10.3390/dj10110206. PMID 36354651
- [Background] Tashbayev B, Rusthen S, Young A, Herlofson BB, Hove LH, Singh PB, Rykke M, Aqrawi LA, Chen X, Utheim OA, Utheim TP, Palm O, Jensen JL. Interdisciplinary, Comprehensive Oral and Ocular Evaluation of Patients with Primary Sjogren's Syndrome. Sci Rep. 2017 Sep 7;7(1):10761. doi: 10.1038/s41598-017-10809-w. PMID 28883442
- See also: The European Code of Conduct for Research Integrity - Revised Edition 2023. Berlin: All European Academies. — https://allea.org/code-of-conduct/
- See also: Asan, M. F., Babu, G. S., Castelino, R. L., Rao, K., & Pandita, V. (2021). Applications of Photobiomodulation Therapy in Oral Medicine-A Review. European Journal of Therapeutics, 27(2), 177-182. https://doi.org/10.5152/eurjther.2021.20080 — https://eurjther.com/index.php/home/article/view/77